CLINICAL TRIAL: NCT06612099
Title: Comparison of the Effects of Aerobic Exercise Training and Mat Pilates Exercise on Blood Pressure, Functional Capacity and Quality of Life in Hypertensive Individuals
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Çağla Yılmaz, Principal Investigator, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21/09/2024-155794
Record Dates: First submitted 2024-09-21; First posted 2024-09-25 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Hypertension
Keywords: Hypertensive Disease; Aerobic exercise; Mat Pilates Exercise; Hypertension; Blood Pressure; Functional capacity; Quality of life (QOL); Physiotherapy and rehabilitation
MeSH Terms: conditions — Hypertension | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Aerobic Exercise Group (Experimental): Individuals in this group will perform aerobic exercise training on a treadmill/bicycle under the supervision of a physiotherapist for a period of 8 weeks, consisting of a total of 24 training sessions. Moderate intensity aerobic exercise training will be set by calculating the target heart rate range. During the training session, individuals will receive a total of 50 minutes of training, consisting of a 10-minute warm-up, 30 minutes of moderate walking/cycling and a 10-minute cool-down period. In addition to the aerobic exercise training group, on the days he does not come to the session, resistance exercises will be taught in the form of 2 sets of 8 repetitions, with weights of 60-80% of 1 maximum repetition, according to the guidelines of the American Sports Medicine Association, and will be given as home exercises.
  Interventions: Other: Aerobic Exercise
- Mat Pilates Exercise Group (Active Comparator): Individuals in this group will perform mat pilates exercises under the supervision of a physiotherapist for a period of 8 weeks, consisting of a total of 24 exercise sessions. During the exercise sessions, individuals will undergo a 50-minute mat pilates exercise program. In addition to the mat pilates exercise group, on the days when he does not come to the session, resistance exercises will be taught in the form of 2 sets of 8 repetitions, 60-80% of 1 maximum repetition, according to the guidelines of the American Sports Medicine Association, and will be given as home exercises.
  Interventions: Other: Mat Pilates Exercise
- Control Group (No Intervention): Hypertensive individuals who meet the inclusion and exclusion criteria will note their blood pressure values 2 days a week for 8 weeks and share them with the physiotherapist. Patients in this group will be instructed to continue their normal lives.

INTERVENTIONS:
Other: Aerobic Exercise — Individuals in this group will perform aerobic exercise training on a treadmill/bicycle under the supervision of a physiotherapist for a period of 8 weeks, consisting of a total of 24 training sessions. Moderate intensity aerobic exercise training will be set by calculating the target heart rate range. During the training session, individuals will receive a total of 50 minutes of training, consisting of a 10-minute warm-up, 30 minutes of moderate walking/cycling and a 10-minute cool-down period. In addition to the aerobic exercise training group, on the days he does not come to the session, resistance exercises will be taught in the form of 2 sets of 8 repetitions, with weights of 60-80% of 1 maximum repetition, according to the guidelines of the American Sports Medicine Association, and will be given as home exercises.
  Arms: Aerobic Exercise Group
Other: Mat Pilates Exercise — Individuals in this group will perform mat pilates exercises under the supervision of a physiotherapist for a period of 8 weeks, consisting of a total of 24 exercise sessions. During the exercise sessions, individuals will undergo a 50-minute mat pilates exercise program. In addition to the mat pilates exercise group, on the days when he does not come to the session, resistance exercises will be taught in the form of 2 sets of 8 repetitions, 60-80% of 1 maximum repetition, according to the guidelines of the American Sports Medicine Association, and will be given as home exercises.
  Arms: Mat Pilates Exercise Group

SUMMARY:
The research aims to compare two different exercise approaches applied to hypertensive individuals. After completion of the research, it will be revealed which exercise approach is more effective on the parameters evaluated in hypertensive individuals. In this context, it is aimed to increase the use of the exercise approach, which is found to be more effective in hypertensive individuals, in the treatment program.

DETAILED DESCRIPTION:
Exercise is an important lifestyle change in treating and controlling hypertension. The International Society of Hypertension recommends increasing physical activity in the long term as a lifestyle intervention to improve blood pressure control and reduce the risk of cardiovascular disease in hypertensive individuals. Regular exercise appears to reduce drug use as part of lifestyle change in the treatment of hypertension. The risk of developing hypertension in individuals with a sedentary lifestyle is higher than in individuals who engage in regular physical activity.

In addition, new exercise programs such as mat pilates exercises are also applied to hypertensive individuals. Mat pilates exercises are a resistance exercise method used worldwide, especially for middle-aged individuals who do not engage in regular physical activity. In addition, Mat pilates exercises have promising effects, reducing short-term systolic blood pressure by 7.4 mmHg and long-term resting systolic blood pressure by 5.8-7.6 mmHg and diastolic blood pressure by 3.3-3.6 mmHg. These data require further research on the use of mat pilates exercises in hypertensive individuals.

The research aims to compare two different exercise approaches applied to hypertensive individuals. After completion of the research, it will be revealed which exercise approach is more effective on the parameters evaluated in hypertensive individuals. In this context, it is aimed to increase the use of the exercise approach, which is found to be more effective in hypertensive individuals, in the treatment program.

ELIGIBILITY:
Inclusion Criteria:

* Hypertension (blood pressure ≥ Individuals diagnosed with 85/135 mmHg) and under medical follow-up,
* Volunteering to participate in the study,
* Not having been included in any exercise program in the last 4 weeks.

Exclusion Criteria:

* Blood pressure Individuals with ≥ 110/180 mmHg,
* Having had a cerebrovascular accident or cardiovascular disease in the last 6 months,
* Having an orthopedic or neurological disorder that prevents walking.
* Having serious cardiovascular/pulmonary disease.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure | 2 months
  During the measurement, the patient should not be talking, should be leaning back, sitting on a chair, without crossing his legs, without crossing his feet, with his feet touching the ground, with his arm supported at heart level, and after resting calmly for at least 5 minutes. After the brachial artery is palpated in the arm, the cuff is placed 2-3 cm below the antecubital fossa. After inflating sufficiently, the pressure will be reduced and the measurement value will be recorded after carefully listening to the beginning and end of the Korotkoff sounds.
Functional Capacity | 2 months
  6 Minute Walk Test will be used to evaluate the submaximal functional capacity of the patients. The aim of this test is to walk the longest distance possible in a 30 meter long corridor within 6 minutes. The testing will be performed in accordance with the guidelines reported by the American Thoracic Society.

SECONDARY OUTCOMES:
Quality of life | 2 months
  The EQ-5D-5L general quality of life scale was developed by the EuroQol group, the Western European Quality of Life Research Society, in 1987 and consists of two parts. The first part is the health profile of that day; It allows it to be defined in five sub-dimensions: movement, self-care, usual activities, pain / discomfort and anxiety / depression. Answers given in each section; It has 5 options: "no problem", "mild problem", "moderate problem", "severe problem" and "extreme problem". The second part consists of the visual analog scale (VAS). In this section, individuals give values between 0 and 100 about their current health status and mark this on a thermometer-like scale. Quality of life scores ranging from 0 to 100 are obtained from the visual analog scale section. As the score of the scale increases, the perception of health increases positively. The Turkish version of the scale, which has been translated into 171 languages by the EuroQol group, will be used in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Çağla Yılmaz, BPT, Principal Investigator — Bezmialem Vakif University; Alis Kostanoğlu, PhD, Study Director — Bezmialem Vakif University; Ahmet Bacaksız, PhD, Study Chair — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Eyüp, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Saco-Ledo G, Valenzuela PL, Ruiz-Hurtado G, Ruilope LM, Lucia A. Exercise Reduces Ambulatory Blood Pressure in Patients With Hypertension: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. J Am Heart Assoc. 2020 Dec 15;9(24):e018487. doi: 10.1161/JAHA.120.018487. Epub 2020 Dec 5. PMID 33280503
- [Background] Ramirez-Jimenez M, Morales-Palomo F, Moreno-Cabanas A, Alvarez-Jimenez L, Ortega JF, Mora-Rodriguez R. Aerobic exercise training improves nocturnal blood pressure dipping in medicated hypertensive individuals. Blood Press Monit. 2022 Aug 1;27(4):272-275. doi: 10.1097/MBP.0000000000000598. Epub 2022 Apr 18. PMID 35438082
- [Background] Caminiti G, Iellamo F, Mancuso A, Cerrito A, Montano M, Manzi V, Volterrani M. Effects of 12 weeks of aerobic versus combined aerobic plus resistance exercise training on short-term blood pressure variability in patients with hypertension. J Appl Physiol (1985). 2021 Apr 1;130(4):1085-1092. doi: 10.1152/japplphysiol.00910.2020. Epub 2021 Feb 25. PMID 33630677
- [Background] Carlin de Ramos do Espirito Santo B, Amante Cardoso L, Sudatti Delevatti R, de la Rocha Freitas C. +Acute blood pressure response after Mat Pilates alone and combined with aerobic exercise. J Bodyw Mov Ther. 2024 Jul;39:579-582. doi: 10.1016/j.jbmt.2024.03.010. Epub 2024 Mar 17. PMID 38876689
- [Background] Martins-Meneses DT, Antunes HK, de Oliveira NR, Medeiros A. Mat Pilates training reduced clinical and ambulatory blood pressure in hypertensive women using antihypertensive medications. Int J Cardiol. 2015 Jan 20;179:262-8. doi: 10.1016/j.ijcard.2014.11.064. Epub 2014 Nov 6. PMID 25464462